CLINICAL TRIAL: NCT01168336
Title: Evaluation of Safety, Drug-Drug Interactions and Pharmacokinetic Profiles of Co-Administration of Escalating Doses of Extended Release and Standard Formulations of Betahistine as Monotherapy and as Adjunctive to Olanzapine in Healthy Subjects
Brief Title: Evaluation of Co-Administration of Betahistine as Adjunctive to Olanzapine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OBEcure Ltd. (Industry)
Responsible Party: Mihaela Pisleaga, PIERREL RESEARCH HP-RO SRL
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: BET 216
Record Dates: First submitted 2010-07-20; First posted 2010-07-23 (Estimated); Last update posted 2010-12-30 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: betahistine olanzapine weight sleepiness; olanzapine induced weight gain and sleepiness
MeSH Terms: conditions — Sleepiness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- betahistine (Experimental): Betahistine 24 mg tablets
  Interventions: Drug: Betahistine standard formulation
- betahistine XR (Experimental): betahistine 32 mg tablets
  Interventions: Drug: Betahistine Extended Release formulation
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Betahistine standard formulation — betahistine 24 mg tablets
  Arms: betahistine
Drug: Betahistine Extended Release formulation — betahistine 32 mg tablets
  Arms: betahistine XR
Drug: Placebo — matching placebo
  Arms: placebo

SUMMARY:
The study aims to evaluate the safety and pharmacokinetics of extended release and standard formulations of betahistine when administered as monotherapy and as compared to their safety and pharmacokinetics when co-administered with olanzapine and to determine potential dose limiting toxicities and/or drug-drug interactions affecting the pharmacokinetics or safety of either medication, with particular emphasis on somnolence and weight gain secondary to olanzapine treatment

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects 18 to 45 years of age and Body Mass Index (BMI)in the range of 18.5 to 27.0
2. Male and females
3. If female - must be non-lactating and non-pregnant, as measured by negative urine pregnancy test, have no plans to become pregnant during the study and practicing appropriate birth control such as oral contraceptives (for at least 60 days ), implants, intrauterine contraceptive devices, sexual abstinence, tubal ligation, or a vasectomized partner, for the study duration
4. Signed written informed consent.
5. Willing and able to comply with study procedures (including reporting to the research center for all weekday evening administrations and staying overnight in the research facility for required PK samplings

Exclusion Criteria:

1. Has a known intolerance, sensitivity or any contraindication to Betahistine or Olanzapine, as delineated in product label
2. Requires chronic or as needed use of systemic antihistamines, anti-obesity agents or psychoactive drugs .
3. Has had a significant body weight loss of over 4 kg in the 90 days prior to screening.
4. Has recently started a smoking cessation program.
5. Has screening ESS score of over 6.
6. Has personal history of gestational diabetes, or has a first degree relative with diabetes.
7. Has any clinically significant abnormality at screening, as judged by Investigator, in laboratory test values (chemistry, hematology, metabolic or urinalysis), including Fasting blood glucose level over 110 mg/dL or HBA1c over 6.0% at screening. Renal insufficiency defined as a serum creatinine over 1.5 mg/dL (133 µmol/L) at screening; Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 ULN; Triglycerides [TG] >200 mg/dL or low-density lipoprotein cholesterol [LDL-C] >190 mg/dL), Thyroid-stimulating hormone (TSH) outside of the normal range;
8. Has any clinically significant abnormality in physical examination or electrocardiogram (ECG), as judged by the Investigator
9. Has a clinically significant history or presence of any disease or unstable medical condition that might be affected by enrollment to this trial, as judged by the Investigator, including; Cardiovascular or cerebrovascular disease Diabetes mellitus (type 1 or 2); Malignant disease within 5 years of screening; Polycystic ovary disease; Hypertension (sitting blood pressure >140/90 mmHg at screening or randomization), History of asthma symptoms in the past 5 years; History of peptic ulcers in the past 5 years; History of HIV, Hepatitis B or Hepatitis C
10. Plans on having any surgery (elective or otherwise) during the course of the study;
11. Has received any investigational drug within 90 days prior to screening.
12. Has been treated over the past 60 days, is currently treated, or is expected to require or undergo treatment with any medications for a period of more than 3 days (with the exception of antibiotic treatment for a period of less than 7 days).
13. Is an immediate family member of personnel directly affiliated with the study at the investigative site, or is personally directly affiliated with the study at the investigative site; or is employed by OBEcure Ltd.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety of escalating doses of extended release and standard formulations of betahistine, as monotherapy and as adjunctive to olanzapine | thisoutcome will be assssed 7 weeks after radomization.
  The total expected duration of the study for each subject will be 7 weeks. Total exposure time to Betahistine alone will be 1 week and total exposure time to Betahistine plus Olanzapine will be 3 weeks.
Evaluation of drug-drug interactions and pharmacokinetic profiles of escalating doses of extended release and standard formulations of betahistine, as adjunctive to olanzapine | 4 weeks
Evaluation of pharmacokinetic profiles of escalating doses of extended release and standard formulations of betahistine, as monotherapy and as adjunctive to olanzapine | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Cinca, Prof MD, Principal Investigator — Pierrel Research HP-RO
Locations (2):
- Romania (2):
  - Pierrel Research HP-RO, Arad
  - Pierrel Research HP-RO, Timișoara